CLINICAL TRIAL: NCT01604291
Title: Multi-Center, Non-Interventional Study, on the Efficacy of Dual and Triple Therapies Based on Pegylated Interferon Alfa-2a for the Treatment of Chronic Hepatitis C Patients
Brief Title: An Observational Study of Dual and Triple Therapies Based on Pegasys (Peginterferon Alfa-2a) in Patients With Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: ML28268
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center, observational study will evaluate the efficacy and safety of dual and triple therapies based on Pegasys (peginterferon alfa-2a) in patients with chronic hepatitis C. Patients receiving treatment with either Pegasys plus ribavirin or Pegasys plus ribavirin plus telaprevir/boceprevir will be observed for the duration of their treatment and for up to 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic hepatitis C (all genotypes, naïve or treatment experienced, HCV mono-infected or HCV-HIV co-infected)
* Receiving either dual therapy (Pegasys plus ribavirin) or triple therapy (Pegasys plus ribavirin plus telaprevir/boceprevir)
* No contra-indications to Pegasys and ribavirin therapy or to treatment regimen containing protease inhibitor (telaprevir or boceprevir) as detailed in local Prescribing Information
* Quantitative serum HCV RNA by PCR test before initiation of treatment

Exclusion Criteria:

* Hepatitis A/B co-infection
* Evidence of severe illness, active malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C patients initiating Pegasys-based treatment
Sampling Method: Probability Sample
Enrollment: 991 (Actual)
Dates: Start 2012-05-28 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2016-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- Israel (21):
  - Haemek Hospital; Gastroenterology, Afula
  - Barzilai MC; Gastroenterology, Ashkelon
  - Soroka Medical Center; Gastroenterology, Beersheba
  - Hillel Yaffe Hospital; Gastroenterology, Hadera
  - Rambam Medical Center; Gastroenterology - Liver Unit, Haifa
  - Bnei-Zion Medical Center; Gastroenterology, Haifa
  - Carmel Hospital; Liver Unit, Haifa
  - Wolfson Hospital; Gastroenterology Unit, Holon
  - Shaare Zedek Hospital Liver Unit; Liver Unit, Jerusalem
  - Hadassah Hospital; Liver Unit, Jerusalem
  - Meir Medical Center; Liver Unit, Kfar Saba
  - Western Galilee Hospital - Nahariya, Nahariya
  - Holy Family Medical Center; Liver Unit, Nazareth
  - Beilinson-Rabin Liver Unit; Liver Unit, Petah Tikva
  - Hasharon Mc; Gastroenterology, Petah Tikva
  - Sheba Medical Center; Tel Hashomer, Ramat Gan
  - Kaplan Medical Center; Gastroenterology Unit, Rehovot
  - Rebecca Sieff Medical Center; Liver Unit, Safed
  - Tel-Aviv Sourasky Medical Center; Liver Unit, Tel Aviv
  - Poria Hospital; Gastroenterology, Tiberias
  - Assaf Harofeh; Gastroenterology, Ẕerifin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 investigational centers in Israel.
Pre-assignment Details: The study was consisted of 3 arms of treatments: 1. Dual therapy: Peginterferon alfa-2a & Ribavirin; 2. Triple therapy :Peginterferon alfa 2a & Ribavirin & Telaprevir; 3. Triple therapy: Peginterferon alfa 2a & Ribavirin & Boceprevir
Groups:
- Peginterferon Alfa-2a + Ribavirin: Dual Therapy. Dosing and treatment duration of the dual therapy (Peginterferon Alfa-2a + Ribavirin) were at the discretion of the Investigator in accordance with the current local prescribing information.
- Peginterferon Alfa-2a + Ribavirin + Telaprevir: Triple Therapy. Dosing and treatment duration of the triple therapy (Peginterferon Alfa-2a + Ribavirin + Teleprevir) were at the discretion of the Investigator in accordance with the current local prescribing information.
- Peginterferon Alfa-2a + Ribavirin + Boceprevir: Triple Therapy. Dosing and treatment duration of the triple therapy (Peginterferon Alfa-2a + Ribavirin + Boceprevir) were at the discretion of the Investigator in accordance with the current local prescribing information.
- No Information on Treatment Allocation: Participants for which Treatment Allocation Data is Unavailable.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2a + Ribavirin + Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir | No Information on Treatment Allocation
Started | 311 | 443 | 193 | 44
Completed | 311 | 443 | 193 | 44
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2a + Ribavirin + Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir | No Information on Treatment Allocation | Total
Number analyzed (Participants) | 311 | 443 | 193 | 44 | 991
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (10.6) | 50.3 (11.0) | 51.1 (11.6) | 48.1 (12.0) | 48.4 (11.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 101 | 161 | 74 | 9 | 345
  Male | 210 | 282 | 118 | 18 | 628
  Unknown | 0 | 0 | 1 | 17 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Viral Response (SVR) at Week 24
Description: The overall SVR-24 rate was defined as percentage of participants with Hepatitis C Virus Ribonucleic Acid (HCV-RNA) levels < 50 International Units per MilliLiter (IU/mL) (as measured by Polymerase Chain Reaction (PCR)) at 24 weeks post treatment completion.
Time Frame: Week 24
Population: Modified All Treated (mTRT) Population: includes all participants who had an HCV-RNA result ≥50 IU/mL at their last measurement prior to commencing CHC therapy; had received one of the study's combination therapies; the participants' treatment documentation was sufficient for assignment to treatment groups.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Peginterferon Alfa-2a + Ribavirin + Telaprevir: Triple Therapy. Dosing and treatment duration of the triple therapy (Peginterferon Alfa-2a + Ribavirin + Telaprevir) were at the discretion of the Investigator in accordance with the current local prescribing information.
- Peginterferon Alfa-2a + Ribavirin + Boceprevir: Triple Therapy. Dosing and treatment duration of the triple therapy (Peginterferon Alfa-2a + Ribavirin +Boceprevir) were at the discretion of the Investigator in accordance with the current local prescribing information.
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2a + Ribavirin + Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 303 | 442 | 190
Percentage of Participants | 87.2 [81.1 to 91.9] | 94.8 [91.6 to 97.1] | 85.2 [77.4 to 91.1]

2. Secondary Outcome: Comparison of SVR at Week 24
Description: SVR at Week 24 is compared by treatment group, type of infection, prior treatments and genotype.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2a + Ribavirin + Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 303 | 442 | 190
Percentage of Participants
  HCV Mono Infection: number analyzed (Participants) | 157 | 287 | 110
  HCV Mono Infection | 86.6 [80.3 to 91.5] | 94.8 [91.5 to 97.0] | 84.5 [77.2 to 91.1]
  HIV/HCV Co-Infection: number analyzed (Participants) | 6 | 5 | 0
  HIV/HCV Co-Infection | 100 [NA to NA] — 100% of participants with HIV/HCV co-infection had a SVR-24 response. | 100 [NA to NA] — 100% of participants with HIV/HCV co-infection had a SVR-24 response. |
  Genotype 1: number analyzed (Participants) | 37 | 292 | 109
  Genotype 1 | 83.8 [68.0 to 93.8] | 94.9 [91.6 to 97.1] | 84.4 [77.2 to 91.1]
  Other Genotypes: number analyzed (Participants) | 127 | 1 | 0
  Other Genotypes | 88.2 [81.3 to 93.2] | 100 [NA to NA] — 100% of participants in this arm with other genotypes had a SVR rate. |
  Treatment - Naive: number analyzed (Participants) | 146 | 110 | 45
  Treatment - Naive | 89.7 [83.6 to 94.1] | 95.5 [89.5 to 98.5] | 86.7 [73.2 to 94.9]
  Treatment - Experienced: number analyzed (Participants) | 18 | 182 | 65
  Treatment - Experienced | 66.7 [41.0 to 86.7] | 94.5 [90.1 to 97.3] | 83.1 [73.6 to 91.9]

3. Secondary Outcome: Number of Participants With SVR at Week 24 According to the Demographic Characteristics
Description: The overall SVR-24 rate was defined as percentage of participants with Hepatitis C Virus Ribonucleic Acid (HCV-RNA) levels < 50 International Units per MilliLiter (IU/mL) (as measured by Polymerase Chain Reaction (PCR)) at 24 weeks post treatment completion. Number of participants analysed signifies participants who were evaluated for outcome measure. Data for this outcome measure was not summarized for each arm. Hence, data is reported for all participants.
Time Frame: Week 24
Population: Participants who treated for chronic hepatitis C(CHC)with either dual therapy (peginterferon alfa-2a and ribavirin)or triple therapy(peginterferon alfa-2a and ribavirin and telaprevir/boceprevir)for up to 24 weeks thereafter in line with local prescribing information at time of study and for whom demographic baseline characteristics were available.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants who had dual or triple therapy as part of their drug regimen at the discretion of the investigator in accordance with the local prescribing information at the time of the study.
Arm/Group | All Participants
Number analyzed (Participants) | 567
Participants
  Gender: Male - Achieved SVR 24 | 316
  Gender: Male - Did not achieve SVR | 33
  Gender: Female - Achieved SVR 24 | 198
  Gender: Female - Did not achieve SVR | 20
  Age - Achieved SVR 24 | 513
  Age - Did not achieve SVR: number analyzed (Participants) | 53
  Age - Did not achieve SVR | 44
  Height - Achieved SVR 24 | 44
  Height - Did not achieve SVR | 44
  Weight - Achieved SVR 24 | 44
  Weight - Did not achieve SVR | 44
  Body Mass Index - Achieved SVR 24 | 44
  Body Mass Index - Did not achieve SVR | 44
Statistical Analysis 1: Comparison: All Participants; Correlation between SVR 24 and Gender; Test type: Other; p = 0.9109, Chi-squared — The p-value from chi-square is the difference between SVR achieved (yes/no) and dose modifications
Statistical Analysis 2: Comparison: All Participants; Correlation between SVR 24 and Age; Test type: Other; p = 0.1163, t-test, 1 sided — A t-test was done to compare SVR participants to non-SVR
Statistical Analysis 3: Comparison: All Participants; Correlation between SVR 24 and Height; Test type: Other; p = 0.9269, t-test, 1 sided — A t-test was done to compare SVR participants to non-SVR
Statistical Analysis 4: Comparison: All Participants; Correlation between SVR 24 and Weight; Test type: Other; p = 0.3376, t-test, 1 sided — A t-test was done to compare SVR participants to non-SVR
Statistical Analysis 5: Comparison: All Participants; Correlation between SVR 24 and Body mass index; Test type: Other; p = 0.4618, t-test, 1 sided — A t-test was done to compare SVR participants to non-SVR

4. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR) at Week 4
Description: RVR was defined as HCV-RNA <50 IU/mL by Week 4
Time Frame: Week 4
Population: mTRT population: participants who had an HCV-RNA result ≥50 IU/mL at their last measurement prior to commencing CHC therapy; had received one of the study's combination therapies; participants' treatment documentation was sufficient for assignment to treatment groups. Number of participants analyzed: participants evaluated for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Peginterferon Alfa-2a + Ribvavirin: Dual Therapy. Dosing and treatment duration of the dual therapy (Peginterferon Alfa-2a + Ribavirin) were at the discretion of the Investigator in accordance with the current local prescribing information.
- Peginterferon Alfa-2a + Ribavirin +Telaprevir: Triple Therapy. Dosing and treatment duration of the triple therapy (Peginterferon Alfa-2a + Ribavirin +Telaprevir) were at the discretion of the Investigator in accordance with the current local prescribing information
Arm/Group | Peginterferon Alfa-2a + Ribvavirin | Peginterferon Alfa-2a + Ribavirin +Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 224 | 398 | 156
Percentage of Participants | 61.2 [54.4 to 67.6] | 70.9 [66.1 to 75.3] | 21.1 [15.0 to 28.4]

5. Secondary Outcome: Percentage of Participants With Extended RVR
Description: Extended RVR was defined as HCV-RNA <50 IU/mL at weeks 4 and 12 for participants treated with telaprevir; or at weeks 8 & 24 for participants treated with boceprevir.
  The assessment was performed in participants who received triple therapy in treatment arms 'Peginterferon Alfa-2a + Ribavirin +Telaprevir' and 'Peginterferon Alfa-2a + Ribavirin + Boceprevir'.
Time Frame: Week 4 and 12 for telaprevir group; Week 8 and 24 for boceprevir group
Population: mTRT population:participants who had an HCV-RNA result ≥50 IU/mL at their last measurement prior to commencing CHC therapy;had received one of study's triple combination therapies;participants' treatment documentation was sufficient for assignment to treatment groups.Number of participants analyzed:participants evaluated for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin +Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 355 | 99
Percentage of Participants | 72.7 [67.7 to 77.2] | 70.7 [60.7 to 79.4]

6. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR)
Description: Complete early virologic response (cEVR) was defined as HCV-RNA <50 IU/mL by Week 12
Time Frame: Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peginterferon Alfa-2a + Ribvavirin | Peginterferon Alfa-2a + Ribavirin +Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 192 | 372 | 158
Percentage of Participants | 75.0 [68.3 to 81.0] | 84.9 [80.9 to 88.4] | 62.0 [54.0 to 69.6]

7. Secondary Outcome: Percentage of Participants With End of Treatment Response (EoT)
Description: End-of-Treatment (EoT) response was defined as HCV-RNA <50 IU/mL by the end of treatment.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peginterferon Alfa-2a + Ribvavirin | Peginterferon Alfa-2a + Ribavirin +Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 286 | 430 | 188
Percentage of Participants | 86.4 [81.8 to 90.1] | 81.9 [77.9 to 85.4] | 76.6 [69.9 to 82.4]

8. Secondary Outcome: Percentage of Participants With Virologic Relapse
Description: Virologic relapse was defined as detectable HCV-RNA during the treatment-free follow-up period in participants with HCV-RNA <50 IU/mL at EoT.
Time Frame: Week 72
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peginterferon Alfa-2a + Ribvavirin | Peginterferon Alfa-2a + Ribavirin +Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 286 | 431 | 188
Percentage of Participants | 0.3 [0 to 1.9] | 0 [NA to NA] — No participants in this arm suffered a virologic relapse. | 0 [NA to NA] — No participants in this arm suffered a virologic relapse.

9. Secondary Outcome: Treatment Duration
Description: The average amount of time a treatment was prescribed to participants.
Time Frame: Week 48
Population: All Enrolled Participants
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2a + Ribavirin + Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 311 | 443 | 193
Weeks
  Peginterferon Alfa-2a Treatment Duration | 26.2 (11.5) | 34.8 (15.2) | 36.1 (14.7)
  Ribavirin Treatment Duration | 26.2 (11.6) | 34.8 (15.2) | 36.1 (14.7)
  Telaprevir/ Boceprevir Treatment Duration | NA (NA) — Participants in this arm did not receive Telaprevir or Boceprevir | 11.8 (4.6) | 30.6 (14.9)

10. Secondary Outcome: Time to First Dose Modification of Peginterferon Alfa-2a
Time Frame: Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2a + Ribavirin +Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 227 | 421 | 187
Days | 418.5 (9.7) | 247.6 (4.1) | 328.4 (13.7)

11. Secondary Outcome: Time to First Dose Modification of Ribavirin
Time Frame: Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Peginterferon Alfa-2a + Ribvavirin | Peginterferon Alfa-2a + Ribavirin +Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 280 | 168 | 109
Days | NA (NA) — No participants in this arm had their Ribavirin dose modified. | 61.4 (3.6) | 89.4 (6.8)

12. Secondary Outcome: Time to First Dose Modification of Telaprevir/Boceprevir
Time Frame: Week 48
Population: mTRT population:participants who had an HCV-RNA result ≥50 IU/mL at their last measurement prior to commencing CHC therapy;had received 1 of study's triple combination therapies;participants' treatment documentation was sufficient for assignment to treatment groups.Number of participants analyzed:participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Peginterferon Alfa-2a + Ribavirin +Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 416 | 181
Days | 124.6 (0.7) | 82.3 (0.8)

13. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  Safety analysis included 2 additional participants in arm 'Peginterferon Alfa-2a + Ribavirin + Telaprevir'. The safety parameters were analyzed by the treatment actually received by the participants.
Time Frame: Week 48
Population: Safety Population. Included only participants who had received at least one dose of peginterferon alfa-2a plus ribavirin or peginterferon alfa-2a plus ribavirin plus telaprevir/boceprevir and had at least one post-baseline safety assessment.
Measure: Number; unit: Percentage of Participants
Groups:
- Peginterferon Alfa-2a + Ribavirin + Telaprevir: Triple Therapy. Dosing and treatment duration of the triple therapy (Peginterferon Alfa-2a + Ribavirin +Telaprevir) were at the discretion of the Investigator in accordance with the current local prescribing information.
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2a + Ribavirin + Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 311 | 445 | 192
Percentage of Participants | 68.8 | 79.3 | 85.9

14. Secondary Outcome: Mean Value of Hemoglobin in Participants With Treatment-Induced Anemia
Time Frame: Week 48
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Grams per Deciliter (g/dl)
Groups:
- Peginterferon Alfa-2a +Ribavirin + Boceprevir: Triple Therapy. Dosing and treatment duration of the triple therapy (Peginterferon Alfa-2a + Ribavirin + Boceprevir) were at the discretion of the Investigator in accordance with the current local prescribing information.
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2a + Ribavirin + Telaprevir | Peginterferon Alfa-2a +Ribavirin + Boceprevir
Number analyzed (Participants) | 78 | 348 | 219
Grams per Deciliter (g/dl) | 9.3 (1.6) | 9.2 (1.3) | 9.5 (1.3)

15. Secondary Outcome: Percentage of Participants With Treatment Regimen for HCV Treatment Induced Anemia
Time Frame: Week 48
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | Peginterferon Alfa-2a + Ribvavirin | Peginterferon Alfa-2a + Ribavirin +Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Number analyzed (Participants) | 78 | 348 | 219
Percentage of Participants
  RVB Dose Reduction | 37 | 56.5 | 53.6
  RBV Temporary Interrupted | 2.5 | 4.5 | 2.3
  RBV Permanently Interrupted | 0 | 1.4 | 0.9
  Use of Erythropotin | 18.5 | 27.3 | 29.1
  Blood Transfusion | 17.3 | 18.8 | 12.7
  DAA Permanently Discontinued | 0 | 1.4 | 0.5
  Peg-IFN a-2a Dose Reduction | 2.5 | 1.1 | 5.5
  No Other Action Done | 32.1 | 22.2 | 25.5
  Other | 6.2 | 4.8 | 2.7

16. Secondary Outcome: Percentage of Participants Who Had SVR at Week 24 With Dose Modifications
Description: Participants with dose modifications who had achieved SVR at Week 24 were reported. Data was collected for all participants who had dose modification of Peginterferon alfa-2a, Ribavirin or Telaprevir/boceprevir in any of the treatment regimen during the study.
Time Frame: Week 24
Population: mTRT population: includes all participants who had an HCV-RNA result ≥50 IU/mL at their last measurement prior to commencing CHC therapy; had received one of the study's combination therapies; the participants' treatment documentation was sufficient for assignment to treatment groups.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 935
percentage of participants
  Peginterferon alfa-2a: number analyzed (Participants) | 435
  Peginterferon alfa-2a | 15.70
  Ribavirin: number analyzed (Participants) | 324
  Ribavirin | 55.56
  Telaprevir/boceprevir: number analyzed (Participants) | 516
  Telaprevir/boceprevir | 0.78
Statistical Analysis 1: Comparison: All Participants; Correlation with dose modification for Peginterferon alfa-2a; Test type: Other; p = 0.0463, Chi-squared; The p-value from chi-square is the difference between SVR achieved (yes/no) and dose modifications; phi-coefficient = -0.0835 — phi-coefficient is a measure of the degree of association between two binary variables
Statistical Analysis 2: Comparison: All Participants; Correlation with dose modification for Ribavirin; Test type: Other; p = 0.2052, Chi-squared; The p-value from chi-square is the difference between SVR achieved (yes/no) and dose modifications; phi-coefficient = 0.0666 — phi-coefficient is a measure of the degree of association between two binary variables
Statistical Analysis 3: Comparison: All Participants; Correlation with dose modification for Telaprevir/boceprevir; Test type: Other; p = 0.0033, Fisher Exact; The p-value from chi-square is the difference between SVR achieved (yes/no) and dose modifications; phi-coefficient = -0.1672 — phi-coefficient is a measure of the degree of association between two binary variables

ADVERSE EVENTS:
Time Frame: Week 48
Description: The Safety Analysis population was defined to include only participants who had received at least one dose of a peginterferon alfa-2a plus ribavirin, or a peginterferon alfa-2a plus ribavirin plus telaprevir/boceprevir and had at least one post-baseline safety assessment. Safety analysis included 2 additional participants in arm 'Peginterferon Alfa-2a + Ribavirin + Telaprevir'. The safety parameters were analyzed by the treatment actually received by the participants.
Groups:
- Peginterferon Alfa-2a + Ribavirin +Telaprevir: Triple Therapy. Dosing and treatment duration of the triple therapy (Peginterferon Alfa-2a + Ribavirin + Teleprevir) were at the discretion of the Investigator in accordance with the current local prescribing information.
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2a + Ribavirin +Telaprevir | Peginterferon Alfa-2a + Ribavirin + Boceprevir
Serious Adverse Events (participants affected / at risk) | 24/311 | 78/445 | 26/192
Other Adverse Events (participants affected / at risk) | 208/311 | 338/445 | 161/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Ribavirin (N=311) | Peginterferon Alfa-2a + Ribavirin +Telaprevir (N=445) | Peginterferon Alfa-2a + Ribavirin + Boceprevir (N=192)
Anaemia (Blood and lymphatic system disorders) | 2 | 30 | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Hearing Impaired (Ear and labyrinth disorders) | 0 | 1 | 0
Diabetes Mellitus (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Papilloedema (Eye disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 5 | 0
Chest Pain (General disorders) | 2 | 1 | 3
Death (General disorders) | 4 | 1 | 0
Face Oedema (General disorders) | 0 | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 5 | 12 | 4
Biliary Colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 2
Cryptococcal Fungaemia (Infections and infestations) | 0 | 1 | 0
Diabetic Foot Infection (Infections and infestations) | 0 | 0 | 1
Ear Infection (Infections and infestations) | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 3
Salmonella Bacteraemia (Infections and infestations) | 0 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gout (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 4 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 1
Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 0
Major Depression (Psychiatric disorders) | 0 | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 1
Calculus Urethal (Renal and urinary disorders) | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1
Renal Colic (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0
Testicular Pain (Reproductive system and breast disorders) | 0 | 1 | 0
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 8 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Renal Stone Removal (Surgical and medical procedures) | 1 | 0 | 0
Vena Cava Filter Removal (Surgical and medical procedures) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Ribavirin (N=311) | Peginterferon Alfa-2a + Ribavirin +Telaprevir (N=445) | Peginterferon Alfa-2a + Ribavirin + Boceprevir (N=192)
Anemia (Blood and lymphatic system disorders) | 44 | 162 | 96
Leukopenia (Blood and lymphatic system disorders) | 16 | 22 | 15
Neutropenia (Blood and lymphatic system disorders) | 27 | 33 | 40
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 43 | 24
Vertigo (Ear and labyrinth disorders) | 23 | 29 | 16
Abdominal Pain (Gastrointestinal disorders) | 16 | 28 | 14
Anorectal Discomfort (Gastrointestinal disorders) | 0 | 27 | 2
Constipation (Gastrointestinal disorders) | 12 | 22 | 12
Diarrhoea (Gastrointestinal disorders) | 17 | 31 | 24
Nausea (Gastrointestinal disorders) | 40 | 59 | 34
Proctalgia (Gastrointestinal disorders) | 6 | 27 | 8
Vomiting (Gastrointestinal disorders) | 17 | 25 | 12
Asthenia (General disorders) | 116 | 169 | 85
Pallor (General disorders) | 5 | 24 | 13
Pyrexia (General disorders) | 47 | 60 | 44
Weight Decreased (Investigations) | 29 | 40 | 14
Decreased Appetite (Metabolism and nutrition disorders) | 51 | 66 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 26 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 25 | 26 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 29 | 37 | 23
Dizziness (Nervous system disorders) | 8 | 23 | 9
Dysgeusia (Nervous system disorders) | 23 | 32 | 42
Headache (Nervous system disorders) | 55 | 49 | 26
Depressed Mood (Psychiatric disorders) | 33 | 32 | 14
Insomnia (Psychiatric disorders) | 20 | 18 | 10
Nervousness (Psychiatric disorders) | 48 | 34 | 16
Sleep Disorder (Psychiatric disorders) | 31 | 27 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 46 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 28 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 39 | 19
Dry Skin (Skin and subcutaneous tissue disorders) | 16 | 25 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 41 | 133 | 44
Rash (Skin and subcutaneous tissue disorders) | 43 | 124 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.